CLINICAL TRIAL: NCT02610101
Title: A Blinded, Nutritional Therapy Study, Using a Modified Specific Carbohydrate Diet in Pediatric Crohn's Disease
Brief Title: Nutritional Therapy Study in Pediatric Crohn's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, David Suskind, Professor of Pediatrics, Seattle Children's Hospital
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB#15606
Record Dates: First submitted 2015-11-16; First posted 2015-11-20 (Estimated); Last update posted 2019-05-24 (Actual); Status verified 2019-04

CONDITIONS: Crohn's Disease
Keywords: Specific Carbohydrate Diet; Diet; Nutrition
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Traditional SCD Diet (Active Comparator): 7 subjects will be randomized to a traditional SCD diet
  Interventions: Other: Traditional SCD Diet
- Modified SCD Diet (Active Comparator): 7 subjects will be randomized to a "modified SCD diet", which includes oatmeal and rice
  Interventions: Other: Modified SCD Diet
- Whole Foods Diet (Active Comparator): 7 subjects will be randomized to a" Whole foods diet" without added sugars
  Interventions: Other: Whole foods diet

INTERVENTIONS:
Other: Traditional SCD Diet — Traditional SCD includes removal of all processed foods as well as all grains, sweetners except for honey and all diary except for yogurt fermented for over 24hrs and some hard cheeses
  Other Names: SCD
  Arms: Traditional SCD Diet
Other: Modified SCD Diet — Food components of the traditional SCD with the addition of rice and oats.
  Other Names: Modified SCD
  Arms: Modified SCD Diet
Other: Whole foods diet — A whole foods diet with removal of processed foods. Removal of corn, wheat, sugar and milk are also apart of this dietary regime.
  Arms: Whole Foods Diet

SUMMARY:
The investigators are doing this research study to answer questions about a nutritional therapy called the Specific Carbohydrate Diet (SCD) for children with active Crohn's Disease (CD). The SCDiet is a diet where all grains such as wheat, barley, corn, rice are restricted. Most dairy products (except certain yogurt) are also restricted. The diet mainly consists of meat, fruits, vegetables, nuts, oils and honey, and is offered to individuals with active Crohn's disease as part of standard of care at Seattle Children's.

For this study, the investigators will have three different dietary groups:

1. Traditional SCD diet group
2. Modified SCD to include oatmeal and rice
3. SCD with whole foods without added sugar

Specifically, the investigators want to know:

* Is the SCD well tolerated?
* Is SCD effective for the treatment for active Crohn's Disease?
* Will the results from the varied three dietary groups have the same results for each patient?

DETAILED DESCRIPTION:
21 patients with CD , mild or moderate disease activity as defined by Pediatric Crohn's disease activity index (PCDAI score of 10-45 ) aged 8 -21 years will enroll into this study.Patient's will be randomized to treatment groups. The treatments for this study will be the:(1) Standard SCD as defined by Elaine Gottschall's Breaking the vicious cycle (2) Modified SCD with added oats and rice (3) Whole foods diet without added sugars. Each patient will receive an initial evaluation including a physical exam, medication review, nutritional guidance and post treatment evaluations.

Initial evaluation: Study subject recipient will have the following lab tests including CBC with differential & platelets, a c-reactive protein, sedimentation rate, an albumin, vitamin D level,Cholesterol, Vitamin A, Vitamin E, Zinc, Folate, a stool study for c. difficile, for bacterial culture and ova and parasite, stool calprotectin and microbiome. Additionally, the investigators will complete a physical exam and document their current medications. The study nutritionist will complete a thorough diet history.

Treatment: Patient's will be randomized to treatment groups. The treatments for this study will be the:(1) Standard SCD as defined by Elaine Gottschall's Breaking the vicious cycle (2) Modified SCD with added oats and rice (3) Whole foods diet without added sugars Families will be given a list of "safe foods" that the patient can eat no matter which group the patient is in. Food will be prepared by a Chef knowledgeable in the SCD and whole food diets. Recipes will be predetermined and families will be able to decide food for patient based upon menus. Patients will receive one-on-one guidance by a Seattle Children's Dietician trained in the SCD during each visit. Prior to each visit patient will fill out a 3 day nutrition log which will be reviewed by the dietician during the clinic visit.

Follow-up: Each study subject will have clinical follow-up at 2 weeks, 4 weeks, 8 weeks and 12weeks. Standardized questionnaires, including the Pediatric Crohn's disease activity index (PCDAI) will be completed during each study visit. Information about tabulating the PCDAI scores, is listed in Appendix A. In addition patients will have a physical exam and standard blood work including CBC, sedimentation rate, C-reactive protein, albumin and stool for microbiome analysis at each follow up visit. This stool will be sent to the University of Washington (Dr. Sam Miller's lab) for analysis;additional stool samples will be sent to Katrine Whitson at UC Irvine for protein analysis. Stool calprotectin will additionally be done at week 4 and 12. Vitamin D level will be measured at week 12. Finally, all patients will meet with the nutritionist at each visit who will complete a thorough diet review. Any questions about the SCD will be addressed at each visit.

All study related information will be stored in the RedCap database. Participant data for the study will be stored electronically in the REDCap platform. The REDCap platform is managed by the Institute for Clinical and Translational Science at the University of Washington. Only IRB approved research team members will have access to the REDCap data platform. Each team member will be granted access to the REDCap data system through a secure login. The information about each participant will be de-identified using a unique study code. Some personal information such as date of birth will be stored in RedCap.

Microbiome:

Some stool from the participants at screening, week 2, 4, 8 and 12 will be stored for microbiome analysis. The samples will be stored at Seattle Children's Hospital in the Clinical Research Center lab in the -80 freezer. These samples will be sent to the University of Washington for microbiome analysis and storage on an as necessary basis. Each of these samples will be de-identified and labeled with a unique study code and visit number. Consent for storage will be part of the Informed Consent process.

ELIGIBILITY:
Inclusion Criteria:

1. Children and adolescents 8 to 21 years old
2. Diagnosis of Crohn's Disease made by a primary gastroenterologist based upon history, physical exam, laboratory/radiological studies and gastrointestinal histology
3. Mild or moderate disease activity based upon PCDAI score (10-45)
4. Parent/guardian and child must be able to comprehend the consent and assent
5. Parent/guardian and participant must be able to attend study visits at baseline, and weeks +2, +4, +8, +12.
6. Patient must not have medication changes for his/her inflammatory bowel disease medications for at least 1 months, unless medically necessary.

Exclusion Criteria:

1. Severe disease with PCDAI >45
2. Active or history of intra abdominal abscess, intra abdominal fistula, stricturing Crohn's disease
3. Other serious medical conditions such as neurological, liver, kidney, autoimmune or systemic disease.
4. Has begun TNF inhibitors within two months prior to study
5. Has had change of maintenance medication within the last month
6. Tobacco, alcohol or illicit drug abuse
7. Pregnant subject recipients will be excluded

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Actual)
Dates: Start 2015-11; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Change in Pediatric Crohn's Disease Activity Index | 12 weeks
  Activity Index is a validated form of measurement for disease activity

SECONDARY OUTCOMES:
Fecal Microbiome Analysis | 12 weeks
  Changes in fecal microbiome as defined by species types and percent of total microbiome will be measured using Metagenomic Phylogenetic Analysis (MetaPhlAn)
Change in C-reactive protein at Baseline and 12 weeks | 12 weeks
  Decrease in C-reactive protein (CRP) by Immunorate by Vitros 4600
Change in Calprotectin at Baseline and 12 weeks | 12 weeks
  Decrease in fecal calprotectin by ELISA

CONTACTS AND LOCATIONS:
Overall Officials: David L Suskind, MD, Principal Investigator — Seattle Children's Hospital and The University of Washington
Locations (1):
- Seattle Children's Hospital, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No
Undecided

REFERENCES:
- [Background] Suskind DL, Wahbeh G, Gregory N, Vendettuoli H, Christie D. Nutritional therapy in pediatric Crohn disease: the specific carbohydrate diet. J Pediatr Gastroenterol Nutr. 2014 Jan;58(1):87-91. doi: 10.1097/MPG.0000000000000103. PMID 24048168